CLINICAL TRIAL: NCT02284087
Title: Assessment of Paired Associative Stimulation Protocols Using Cerebellar or Visual Afferences in Post-stroke Hand Motor Deficits
Brief Title: Paired Associative Stimulation in Post-stroke Hand Motor Deficits
Acronym: PAS-stroke
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C14-38; 2014-A01165-42 (Registry Identifier: IDBRCB)
Record Dates: First submitted 2014-10-21; First posted 2014-11-05 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Stroke and Healthy Subjects
Keywords: transcranial magnetic stimulation; movement disorders
MeSH Terms: conditions — Stroke; Movement Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- V_PAS: Visuomotor paired associative stimulation protocol
  Interventions: Device: PAS
- Sham V_PAS: Placebo group of Visuomotor paired associative stimulation protocol
- CER_PAS: cerebellar-motor associative stimulation protocol
  Interventions: Device: PAS
- Sham CER_PAS: Placebo group of cerebellar-motor associative stimulation protocol

INTERVENTIONS:
Device: PAS
  Groups: CER_PAS; V_PAS

SUMMARY:
Introduction The motor impairment of the upper extremity is the most common sequelae after ischemic stroke. Transcranial magnetic stimulation (TMS) is a promising non- invasive technique in the rehabilitation of motor deficits. However, its effect in post-stroke motor deficits remains moderate our days. To potentiate the effect of TMS, techniques called Paired Associative Stimulations (PAS) involving the integration of afferent sensory inputs at the level of the ipsilesional primary motor cortex were developed in healthy subjects. PAS techniques have shown a gain of corticospinal excitability by such phenomenon known as long Term Potentiation (LTP) and a gain of motor performance. The investigators would like to propose to evaluate two types of these techniques with a volley of visual afferents (visuomotor stimulation, V_PAS) or of cerebellar afferents (CER_PAS), because these two structures convey important information in the execution of the movement.

Design Multicenter, randomized, study, 60 patients in 3 parallel groups (V_PAS, CER_PAS, control group with sham and sham V_PAS CER_PAS), 5 days of treatment, clinical assessment, electrophysiological and MRI before, immediately post- and second post-assessments (4 weeks).

A group of 24 healthy subjects will undergo a parallel physiopathological study on the underlying mechanisms of cerebellar PAS

Objectives Main objective: To determine whether (and how) Paired Associative Stimulation technique (PAS) induces cerebral reorganization in the primary motor cortex compared to the control group.

Aim 2: Determine whether (and which) type of PAS is capable of inducing changes in motor performance of the upper limb paresis and duration Aim 3: Determine whether (and which) type of PAS is capable of inducing changes in excitability of the corticospinal tract and duration Aim 4: Determine how PAS techniques modify the functional connectivity during movement Aim 5: Determine if connectivity changes during induced movement correlate with clinical improvements Aim 6: Determine whether patients who benefit of a type of PAS have specific anatomical lesion characteristics (volume, afferent and efferent white matter fasciculi integrity)

DETAILED DESCRIPTION:
Introduction The motor impairment of the upper extremity is the most common sequelae after ischemic stroke. Transcranial magnetic stimulation (TMS) is a promising non- invasive technique in the rehabilitation of motor deficits. However, its effect in post-stroke motor deficits remains moderate the investigators days. To potentiate the effect of TMS, techniques called Paired Associative Stimulations (PAS) involving the integration of afferent sensory inputs at the level of the ipsilesional primary motor cortex were developed in healthy subjects. PAS techniques have shown a gain of corticospinal excitability by such phenomenon known as long Term Potentiation (LTP) and a gain of motor performance. The investigators would like to propose to evaluate two types of these techniques with a volley of visual afferents (visuomotor stimulation, V_PAS) or of cerebellar afferents (CER_PAS), because these two structures convey important information in the execution of the movement.

Design Multicenter, randomized study, 60 patients in 3 parallel groups (V_PAS, CER_PAS, control group with sham and sham V_PAS CER_PAS), 5 days of treatment, clinical assessment, electrophysiological and MRI before, immediately post- and second post-assessments (4 weeks).

A group of 24 healthy subjects will undergo a parallel physiopathological study on the underlying mechanisms of cerebellar PAS Objectives Main objective: To determine whether (and how) Paired Associative Stimulation technique (PAS) induces cerebral reorganization in the primary motor cortex compared to the control group.

Aim 2: Determine whether (and which) type of PAS is capable of inducing changes in motor performance of the upper limb paresis and duration Aim 3: Determine whether (and which) type of PAS is capable of inducing changes in excitability of the corticospinal tract and duration Aim 4: Determine how PAS techniques modify the functional connectivity during movement Aim 5: Determine if connectivity changes during induced movement correlate with clinical improvements Aim 6: Determine whether patients who benefit of a type of PAS have specific anatomical lesion characteristics (volume, afferent and efferent white matter fasciculi integrity) Aim 7: for healthy subjects: determine the TMS parameters that will influence the response to cerebellar PAS protocols

Hypotheses

* The sensorimotor stimulation approach (V_PAS or CER_PAS) improves motor function of the hand compared to the control group. The CER_PAS approach may be more effective than V_PAS as the cerebellum plays a major role in the post-stroke recovery
* This improvement would be explained by an effect on brain reorganization by increasing the proportion of activation in the ipsilesional primary motor cortex comparing to the contralesional side, as well as strengthening the relationships between ipsilesional premotor and motor cortices.
* Clinical and electrophysiological effects observed in the combined approach are correlated with specific characteristics of the sensorimotor network assessed by MRI.

Perspectives Demonstrating beneficial effects would subsequently consider protocols in order to achieve a therapeutic effect in the long term. The low cost greatly facilitates the implementation of feasible treatments in routine care in specialized centers (or pilot research centers) and potentially useful in many patients. The study of the characteristics of responders and non-responders patients would provide "patient-oriented" treatment, which take into account the particularities of each subject.

ELIGIBILITY:
Inclusion Criteria FOR PATIENTS:

* First event ischemic stroke with hand motor deficit
* Time since stroke > 30 days
* Stroke lesion sparing the primary motor cortex (hand knob area)
* Age between 18 and 85 ans

Exclusion Criteria FOR PATIENTS:

* No homonymous hemianopia
* No contra-indications for TMS and MRI
* Pregnancy
* Epilepsia
* Any pathology that threatened the 1 month follow up

Inclusion Criteria FOR HEALTHY SUBJECTS:

* Age between 18 and 85
* Right handed

Exclusion Criteria FOR HEALTHY SUBJECTS

* No contra-indications for TMS and MRI
* Pregnancy
* Any cerebral pathology or pathology that threatened the 1 month follow up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
change in lateralization indices in the primary motor cortex using functional magnetic Resonance | Change from Baseline to day 5 (Pre and post intervention)

SECONDARY OUTCOMES:
change in motor score of the affected hand by the Jebsen Taylor Test | Change from Baseline to day 5 (Pre and post intervention)
change in corticospinal excitability by the motor evoked potentials | Change from Baseline to day 5 (Pre and post intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte ROSSO, PI, Principal Investigator — Brain and Spine institute, INSERM UMR 1127, CNRS 7225
Locations (1):
- ICM, CIC Neurosciences, Paris, France

REFERENCES:
- [Result] Rosso C, Moulton EJ, Kemlin C, Leder S, Corvol JC, Mehdi S, Obadia MA, Obadia M, Yger M, Meseguer E, Perlbarg V, Valabregue R, Magno S, Lindberg P, Meunier S, Lamy JC. Cerebello-Motor Paired Associative Stimulation and Motor Recovery in Stroke: a Randomized, Sham-Controlled, Double-Blind Pilot Trial. Neurotherapeutics. 2022 Mar;19(2):491-500. doi: 10.1007/s13311-022-01205-y. Epub 2022 Feb 28. PMID 35226342
- [Result] Kemlin C, Moulton E, Leder S, Houot M, Meunier S, Rosso C, Lamy JC. Redundancy Among Parameters Describing the Input-Output Relation of Motor Evoked Potentials in Healthy Subjects and Stroke Patients. Front Neurol. 2019 May 21;10:535. doi: 10.3389/fneur.2019.00535. eCollection 2019. PMID 31178817
- [Result] Rosso C, Perlbarg V, Valabregue R, Obadia M, Kemlin-Mechin C, Moulton E, Leder S, Meunier S, Lamy JC. Anatomical and functional correlates of cortical motor threshold of the dominant hand. Brain Stimul. 2017 Sep-Oct;10(5):952-958. doi: 10.1016/j.brs.2017.05.005. Epub 2017 May 17. PMID 28551318
- [Result] Rosso C, Lamy JC. Does Resting Motor Threshold Predict Motor Hand Recovery After Stroke? Front Neurol. 2018 Nov 29;9:1020. doi: 10.3389/fneur.2018.01020. eCollection 2018. PMID 30555404